CLINICAL TRIAL: NCT04027764
Title: Toripalimab Combined With S1 and Albumin Paclitaxel as First Line in Patients With Advanced Biliary Tract Cancer: a Single-arm,One Center， Phase II Clinical Study
Brief Title: Toripalimab Combined With S1 and Albumin Paclitaxel in Patients With Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dai, Guanghai (Other)
Responsible Party: Sponsor-Investigator, Dai, Guanghai, professor,deputy cheif of oncology department, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSA-01
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Advanced Biliary Tract Cancer
Keywords: advanced biliary tract cancer; Albumin Paclitaxel; s1; Toripalimab
MeSH Terms: interventions — S 1 (combination); theasinensin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined With S1 and Albumin Paclitaxel (Experimental)
  Interventions: Drug: Toripalimab Combined With S1 and Albumin Paclitaxel

INTERVENTIONS:
Drug: Toripalimab Combined With S1 and Albumin Paclitaxel — Toripalimab 240 mg ，every 2-3 weeks S1：80-120mg，bid；oral，d1-14； Albumin Paclitaxel：120mg/m2，D 1 \8
  Other Names: TSA

SUMMARY:
The investigator's study is a single armed phrase II trial ,aiming to improve the effecacy of treatment for advanced billiary tract cancer by means of Toripalimab combining with S1 and Albumin Paclitaxel as first line in patients with advanced Biliary Tract Cancer. treatment continually until disease progression or intolerable toxicity or Patients withdrawal of consent.and target sample is 30+ patients.

DETAILED DESCRIPTION:
Toripalimab: 240 mg , once every 2-3 weeks; S1: 80-120mg, bid; oral, day1-14; Albumin paclitaxel: 120mg/m2 , administered on the first day and the eighth day of each cycle; 21 days for a treatment cycle

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients with gallbladder and cholangiocarcinoma diagnosed by histology or cytology
3. Liver function Child-Pugh grade A (5-6 points) or better grade B (≤ 7 points)
4. ECOG score 0 or 1 point
5. At least one measurable lesion
6. no previous treatment

Exclusion Criteria:

1. organs failure ,including liver ,heart ,kidney
2. Have received a liver transplant in the past
3. Active brain metastasis or spinal cord compression
4. ECOG score 3 or 4 point
5. Symptomatic peripheral neuropathy (CTCAE ≥ 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 year
  ORR

SECONDARY OUTCOMES:
progression free survival | 1 year
  PFS
disease response rate | 1 year
  DCR
overall survival | 1 year
  OS

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No